CLINICAL TRIAL: NCT00858156
Title: An Open-Label, Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Oral BG9928 in Subjects With Mild and Moderate Hepatic Impairment and in Healthy Subjects
Brief Title: BG9928 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec, Medical Director, Biogen Idec, Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 161HI101
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Hepatic Impairment
Keywords: Pharmacokinetics
MeSH Terms: interventions — BG 9928

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BG9928 — Oral 75 mg single dose

SUMMARY:
The primary objective of the study is to evaluate the effect of hepatic function on the pharmacokinetics of a single oral dose of BG9928 in subjects with mild and moderate hepatic impairment and in subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 75, inclusive.
* Must have a Body Mass Index (BMI) between 19 kg/m2 and 36 kg/m2, inclusive.

The following criteria apply only to subjects enrolled into Groups 1 and 2 (mild or moderate hepatic impairment):

* Must have stable hepatic disease (i.e., no change in disease status within the last 2 months as determined by the enrolling Investigator) with laboratory and clinical findings that support the diagnosis of hepatic impairment.
* Must have a total Child-Pugh score (Section 22, Appendix I) of 5-6 (mild), or 7-9 (moderate).
* Must be otherwise healthy as determined by the Investigator on the basis of pre-study physical examination, medical history, 12-lead ECG, vital signs, and clinical laboratory parameters. Subjects with controlled hypertension and those problems directly associated with the primary diagnosis of hepatic impairment may be included. Subjects with stable, mild, chronic concurrent diseases, such as degenerative joint disease, may be included.

Exclusion Criteria:

* History of an allergic reaction to any methylxanthine-containing compound.
* History of seizure within the past 10 years, or use of any medication for the suppression of seizures within the past 5 years.
* History of brain surgery, meningitis/encephalitis, penetrating head trauma, stroke, or transient ischemic attack within the past 6 months.
* History of active (within 6 months) drug or alcohol abuse, a positive drug screen (without a medically indicated rationale), or a positive alcohol breath test at Screening or on Day -2.
* History of Human Immunodeficiency Virus (HIV) antibody.
* Serious systemic infection (e.g., septicemia) within the 30 days prior to Day 1.
* Fever, with body temperature >38oC, within the 48 hours prior to Day 1.
* Active bacterial or viral infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The comparative effect of hepatic function on the pharmacokinetics of a single oral dose of BG9928 in subjects with mild and moderate hepatic impairment as compared to subjects with normal hepatic function | 1 week post dose

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec, Study Director — Biogen
Locations (2):
- United States (2):
  - Miami, Florida
  - Orlando, Florida